CLINICAL TRIAL: NCT06136806
Title: Diagnostic Performance of a Novel Ferumoxytol-Enhanced Coronary Magnetic Resonance Angiography/ Venography on Panvascular Disease: a Single-center Clinical Study.
Brief Title: Diagnostic Performance of a Novel Ferumoxytol-Enhanced Magnetic Resonance Angiography/ Venography on Panvascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Chief leader of CCU, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 027
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2023-11

CONDITIONS: Panvascular Disease
Keywords: Magnetic Resonance Imaging; Ferumoxytol; Panvascular Disease
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Multisite Artery Disease (MAD) Group: Participants in MAD group mean these patients are suspected with multisite artery disease, like coronary artery disease accompany with renal artery stenosis or lower extremity atherosclerosis.
  Interventions: Diagnostic Test: Ferumoxytol Enhanced Magnetic Resonance Angiography（ FE-MRA）；Coronary/Renal /Lower artery Arteriography
- Venous Thromboembolism （VTE）Group: Participants in VTE group mean these patients are suspected with deep vein thrombosis or pulmonary embolism.
  Interventions: Diagnostic Test: Ferumoxytol Enhanced Magnetic Resonance Venography（ FE-MRV）, Computed Tomography Pulmonary Angiography, Ultrasound for Lower Extremity Deep Vein.

INTERVENTIONS:
Diagnostic Test: Ferumoxytol Enhanced Magnetic Resonance Angiography（ FE-MRA）；Coronary/Renal /Lower artery Arteriography — When the patient is suspected with multisite artery disease, FE-MRA and angiography will be performed according to the patient's clinical manifestation. For example, when the patient is suspected with coronary artery disease, coronary FE-MRA and angiography will be performed; when the patient is suspected with renal artery stenosis, renal artery FE-MRA and angiography will be performed; and when the patient is suspected with the lower extremity artery occlusion, the lower extremity artery FE-MRA and angiography will be performed.
  Groups: Multisite Artery Disease (MAD) Group
Diagnostic Test: Ferumoxytol Enhanced Magnetic Resonance Venography（ FE-MRV）, Computed Tomography Pulmonary Angiography, Ultrasound for Lower Extremity Deep Vein. — When the patient is suspected with venous thromboembolism, the lower extremity vein FE-MRV, pulmonary FE-MRA and ultrasound for lower extremity deep vein as well as computed tomography pulmonary angiography will be taken to ensure whether the patient with thrombus or not.
  Groups: Venous Thromboembolism （VTE）Group

SUMMARY:
The goal of this observational study is to test the diagnostic performance of ferumoxytol-enhanced magnetic resonance angiography/ venography（FE-MRA/MRV） on panvascular disease. The main questions it aims to answer are:

1. How about the imaging quality of FE-MRA/MRV for panvascular disease?
2. What is the diagnostic performance of FE-MRA/MRV for panvascular disease?

Participants will be divided into two groups based on their symptoms, body signs or laboratory examinations. Participants who suspected with multisite atherosclerotic diseases like coronary artery disease accompany with renal artery stenosis or peripheral arterial disease will be recruited in multisite artery disease (MAD) group. While participants who suspected with venous thromboembolism (VTE) like pulmonary embolism or deep vein thrombosis will be recruited in VTE group. Participants in MAD group will take both FE-MRA and percutaneous selective angiography measurements of coronary, renal, or lower extremity artery, while participant in VTE group need to do pulmonary artery FE-MRA and computed tomography pulmonary angiography (CTPA), lower extremity vein FE-MRV and ultrasonography.

DETAILED DESCRIPTION:
Panvascular disease refers to multi-site vascular disease, presenting as multi-site atherosclerotic disease and venous thromboembolism. There is no gold standard test for panvascular disease up to now. Clinical tests of the suspected population are often carried out by parts and times, and there is no one-stop, panoramic examination on panvascular disease.

Ferumoxytol is a novel and safe MRI contrast agent with an intravascular half-life of approximately 15 hours, enabling simultaneous scanning of multiple sites. At this background, our study intends to investigate the diagnostic efficacy of FE-MRA/MRV in panvascular diseases.

In this study, we plan to enroll 200 patients with suspected panvascular disease. Patients with suspected coronary artery disease, renal artery stenosis, or lower extremity arterial disease will be included in the MAD group, and patients with suspected pulmonary artery embolism and lower extremity venous embolism will be included in the VTE group.

In the MAD group, patients will take both FE-MRA and percutaneous selective angiography of coronary, renal, or lower extremity artery. We will record the FE-MRA image quality score, signal to noise ratio(SNR), compare signal-to-noise ratio（CNR）, whether the coronary, renal, and lower extremity arteries have stenosis greater than 50%, and whether the below-knee arteries are occluded. In the VTE group, patients need to do pulmonary artery FE-MRA and computed tomography pulmonary angiography (CTPA), lower extremity vein FE-MRV and ultrasonography. We will record the image quality scores of FE-MRA of the pulmonary arteries, the FE-MRV the lower extremities, SNR, CNR, the presence of pulmonary embolism or deep vein thrombosis.

The sensitivity, specificity, positive predictive value, and negative predictive value of FE-MRA for the diagnosis of arteries stenosis >50% will be evaluated by using percutaneous selective angiography as the gold standard and generating subject operating characteristic (ROC) curves. And the sensitivity, specificity, positive predictive value, and negative predictive value of FE-MRA/MRV for the diagnosis of thrombosis in the pulmonary artery or lower extremities will be evaluated by generating ROC curves by using CTPA and venous ultrasound as the reference.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years;
2. Those with suspected multi-site atherosclerotic vascular disease (MAD) (fulfilling both a), and at least two of b), c), and d)):

   1. have at least 1 risk factor for atherosclerosis (hypertension, diabetes mellitus, hyperlipidemia, smoking, and obesity);
   2. Those with suspected coronary atherosclerotic cardiovascular disease: angina symptoms, ST-T changes on ECG;
   3. those with suspected atherosclerotic renal artery stenosis: periumbilical vascular murmur, intractable hypertension, renal insufficiency difficult to explain by other causes;
   4. Those with suspected atherosclerotic lower extremity peripheral arterial disease: intermittent claudication, diminished or absent dorsalis pedis arterial pulses.
3. Those with suspected venous thromboembolism (VTE) (fulfill at least one of a) and b)):

   1. Those with suspected DVT: swelling and pain in the lower extremities;
   2. Those with suspected PE: simplified Wells score ≥ 1.
4. Patients sign an informed consent form.

Exclusion Criteria:

1. Those who are allergic to iodine contrast media or have a history of allergy or hypersensitivity to iron or dextrose;
2. Those who are unable to undergo MRI due to psychological (e.g., suffering from claustrophobia syndrome) or physical reasons (e.g., retention of metallic objects in the body);
3. Those with terminal illness (e.g., suffering from malignant tumors) or with a life expectancy of <1 year;
4. Liver insufficiency (alanine aminotransferase > 3 times the upper limit of normal value);
5. Renal insufficiency (eGFR <30mL/min/1.73cm2);
6. Hyperthyroidism;
7. Those with hemodynamic instability;
8. Pregnant and lactating women;
9. Persons with hearing limitations;
10. Persons with cardiac function class III-IV;
11. Persons on other oral or intravenous iron supplements;
12. Patients with ferrous hemosiderin deposition or hemochromatosis;
13. Patients with acute coronary syndromes;
14. Any other person who, in the opinion of the investigator, should not participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study adopts a continuous enrollment method. It is estimated that 200 suspected pan-vascular disease patients will be enrolled within the study period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
the degree of coronary/ renal/lower extremity artery stenosis | 1 week
  Degree of artery stenosis assessed by FE-MRA and percutaneous selective angiography.
Deep Vein Thrombosis | 1 week
  FE-MRV and ultrasound for lower extremity deep vein will be taken to evaluate whether there is deep vein thrombosis or not.
Pulmonary Embolism | 1 week
  FE-MRA and computed tomography pulmonary angiography will be taken to evaluate whether there is pulmonary embolism or not.
Image quality of FE-MRA/MRV | 1 week
  The image quality will be assessed by a 4-point scale:
  1. poor (vessel barely evident or noisy image);
  2. moderate (vessel visible but diagnostic confidence low);
  3. good (vessel adequately visualized and diagnostic quality image);
  4. excellent (vessel clearly depicted)
signal-to-noise ratio （SNR） | 1 week
  An indicator represents for image quality.
contrast-to-noise ratio (CNR) | 1 week
  An indicator represents for image quality.
below-knee artery occlusion | 1 week
  Whether below-knee arteries occlusion or not assessed by FE-MRA and percutaneous selective angiography .

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Esmatjes E, Blanco AJ. [The REACH registry: baseline and 1-year results]. Med Clin (Barc). 2009 Sep;132 Suppl 2:5-9. doi: 10.1016/S0025-7753(09)71745-2. Spanish. PMID 19631831
- [Background] Pan Y, Jing J, Cai X, Jin Z, Wang S, Wang Y, Zeng C, Meng X, Ji J, Li L, Lyu L, Zhang Z, Mei L, Li H, Li S, Wei T, Wang Y. Prevalence and Vascular Distribution of Multiterritorial Atherosclerosis Among Community-Dwelling Adults in Southeast China. JAMA Netw Open. 2022 Jun 1;5(6):e2218307. doi: 10.1001/jamanetworkopen.2022.18307. PMID 35759265
- [Background] Di Noi P, Brancati MF, Burzotta F, Trani C. Multisite artery disease: a common and challenging clinical condition calling for specific management. Future Cardiol. 2014 May;10(3):395-407. doi: 10.2217/fca.14.25. PMID 24976476
- [Background] Zhang Q, Wang A, Zhang S, Li N, Chen S, Zhang Y, Zhou Y, Wu S, Zhao X. Asymptomatic polyvascular disease and the risks of cardiovascular events and all-cause death. Atherosclerosis. 2017 Jul;262:1-7. doi: 10.1016/j.atherosclerosis.2017.04.015. Epub 2017 Apr 21. PMID 28463782
- [Background] Doherty S. Pulmonary embolism An update. Aust Fam Physician. 2017 Nov;46(11):816-820. PMID 29101916
- [Background] Mezquita AJV, Biavati F, Falk V, Alkadhi H, Hajhosseiny R, Maurovich-Horvat P, Manka R, Kozerke S, Stuber M, Derlin T, Channon KM, Isgum I, Coenen A, Foellmer B, Dey D, Volleberg RHJA, Meinel FG, Dweck MR, Piek JJ, van de Hoef T, Landmesser U, Guagliumi G, Giannopoulos AA, Botnar RM, Khamis R, Williams MC, Newby DE, Dewey M. Clinical quantitative coronary artery stenosis and coronary atherosclerosis imaging: a Consensus Statement from the Quantitative Cardiovascular Imaging Study Group. Nat Rev Cardiol. 2023 Oct;20(10):696-714. doi: 10.1038/s41569-023-00880-4. Epub 2023 Jun 5. PMID 37277608
- [Background] Zeng Y, He R, Ren Y, Che Y, Wang G. Cervicocerebral Computed Tomography Angiography for Older Patients Based on Time to Peak and Number of Time Points to Peak in the Test Bolus Technique. J Comput Assist Tomogr. 2023 Jan-Feb 01;47(1):165-172. doi: 10.1097/RCT.0000000000001396. Epub 2022 Dec 13. PMID 36668985
- [Background] Briley-Saebo KC, Cho YS, Shaw PX, Ryu SK, Mani V, Dickson S, Izadmehr E, Green S, Fayad ZA, Tsimikas S. Targeted iron oxide particles for in vivo magnetic resonance detection of atherosclerotic lesions with antibodies directed to oxidation-specific epitopes. J Am Coll Cardiol. 2011 Jan 18;57(3):337-47. doi: 10.1016/j.jacc.2010.09.023. Epub 2010 Nov 23. PMID 21106318
- [Background] Corot C, Robert P, Idee JM, Port M. Recent advances in iron oxide nanocrystal technology for medical imaging. Adv Drug Deliv Rev. 2006 Dec 1;58(14):1471-504. doi: 10.1016/j.addr.2006.09.013. Epub 2006 Sep 30. PMID 17116343
- [Background] Spinowitz BS, Kausz AT, Baptista J, Noble SD, Sothinathan R, Bernardo MV, Brenner L, Pereira BJ. Ferumoxytol for treating iron deficiency anemia in CKD. J Am Soc Nephrol. 2008 Aug;19(8):1599-605. doi: 10.1681/ASN.2007101156. Epub 2008 Jun 4. PMID 18525001
- [Background] Lehrman ED, Plotnik AN, Hope T, Saloner D. Ferumoxytol-enhanced MRI in the peripheral vasculature. Clin Radiol. 2019 Jan;74(1):37-50. doi: 10.1016/j.crad.2018.02.021. Epub 2018 May 3. PMID 29731126
- [Background] Finn JP, Nguyen KL, Hu P. Ferumoxytol vs. Gadolinium agents for contrast-enhanced MRI: Thoughts on evolving indications, risks, and benefits. J Magn Reson Imaging. 2017 Sep;46(3):919-923. doi: 10.1002/jmri.25580. Epub 2017 Feb 3. No abstract available. PMID 28160356
- [Background] Gahramanov S, Raslan AM, Muldoon LL, Hamilton BE, Rooney WD, Varallyay CG, Njus JM, Haluska M, Neuwelt EA. Potential for differentiation of pseudoprogression from true tumor progression with dynamic susceptibility-weighted contrast-enhanced magnetic resonance imaging using ferumoxytol vs. gadoteridol: a pilot study. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):514-23. doi: 10.1016/j.ijrobp.2009.10.072. Epub 2010 Apr 13. PMID 20395065
- [Background] Neuwelt EA, Hamilton BE, Varallyay CG, Rooney WR, Edelman RD, Jacobs PM, Watnick SG. Ultrasmall superparamagnetic iron oxides (USPIOs): a future alternative magnetic resonance (MR) contrast agent for patients at risk for nephrogenic systemic fibrosis (NSF)? Kidney Int. 2009 Mar;75(5):465-74. doi: 10.1038/ki.2008.496. Epub 2008 Oct 8. PMID 18843256
- [Background] Weinstein JS, Varallyay CG, Dosa E, Gahramanov S, Hamilton B, Rooney WD, Muldoon LL, Neuwelt EA. Superparamagnetic iron oxide nanoparticles: diagnostic magnetic resonance imaging and potential therapeutic applications in neurooncology and central nervous system inflammatory pathologies, a review. J Cereb Blood Flow Metab. 2010 Jan;30(1):15-35. doi: 10.1038/jcbfm.2009.192. Epub 2009 Sep 16. PMID 19756021
- [Background] Walker JP, Nosova E, Sigovan M, Rapp J, Grenon MS, Owens CD, Gasper WJ, Saloner DA. Ferumoxytol-enhanced magnetic resonance angiography is a feasible method for the clinical evaluation of lower extremity arterial disease. Ann Vasc Surg. 2015 Jan;29(1):63-8. doi: 10.1016/j.avsg.2014.09.003. Epub 2014 Sep 28. PMID 25269682
- [Background] Dong Z, Si G, Zhu X, Li C, Hua R, Teng J, Zhang W, Xu L, Qian W, Liu B, Wang J, Wang T, Tang Y, Zhao Y, Gong X, Tao Z, Xu Z, Li Y, Chen B, Kong X, Xu Y, Gu N, Li C. Diagnostic Performance and Safety of a Novel Ferumoxytol-Enhanced Coronary Magnetic Resonance Angiography. Circ Cardiovasc Imaging. 2023 Jul;16(7):580-590. doi: 10.1161/CIRCIMAGING.123.015404. Epub 2023 Jul 18. PMID 37463240